CLINICAL TRIAL: NCT01640483
Title: Differential Efficacy of Supportive and Interpretative Psychodynamic Techniques for Dependent and Self-critical Depressive Patients: an Experimental Single Case Design.
Brief Title: Differential Efficacy of Supportive and Interpretative Psychodynamic Techniques for Dependent and Self-critical Depressive Patients
Acronym: PsychodynDep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Funding by BOF (Bijzonder Onderzoeksfonds) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EC/2012/455
Record Dates: First submitted 2012-07-05; First posted 2012-07-13 (Estimated); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- supportive (Active Comparator)
  Interventions: Other: psychodynamic techniques.
- interpretative (Active Comparator)
  Interventions: Other: psychodynamic techniques.
- mixed supportive/interpretative (Active Comparator)
  Interventions: Other: psychodynamic techniques.

INTERVENTIONS:
Other: psychodynamic techniques. — the patients go through a time-limited (50 sessions, 45 minutes, 2 sessions/week) experimental treatment which exists of a sequence of four A phases (control conditions), one B phase (supportive techniques only), one C phase (interpretative techniques only), and one BC phase (mixed supportive/interpretative techniques).

SUMMARY:
Post-hoc analysis of psychotherapy outcome data suggest that psychodynamic techniques for Major Depressive Disorder are differentially efficacious dependent on personality traits of the patient. More specifically, supportive techniques are hypothesized to be more efficacious for dependent patients, interpretative techniques to be more efficacious for self-critical patients, and mixed supportive/interpretative techniques to be more efficacious for mixed dependent/self-critical patients. Moreover, supportive techniques are hypothesized to impact on depressive symptoms through increased relational capacities while interpretative techniques impact through increased self-understanding.

These hypotheses are tested in an experimental single case design with three dependent, three self-critical and three mixed dependent/self-critical depressive patients. These patients go through a time-limited (50 sessions) experimental treatment which exists of a sequence of four A phases (control conditions), one B phase (supportive techniques only), one C phase (interpretative techniques only), and one BC phase (mixed supportive/interpretative techniques).

ELIGIBILITY:
Inclusion Criteria:

* Patient meets criteria for Major Depressive Disorder (as assessed by SCID-I and DSM-IV-TR)
* Patient is prepared to give informed consent

Exclusion Criteria:

* Patient uses antidepressant medication during the treatment
* Patient scores 3 on the suicide item of the BDI-II
* Patient meets criteria for psychotic or personality disorder (as assessed by SCID-II)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2012-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Reduction in depressive symptoms at 25 weeks (50 sessions, 2 sessions/week). | 25 weeks
  •Measures each session: The BDI-II with adapted instructions is used to measure depressive symptoms. The process variables associated with change in depressive symptoms will be studied in an exploratory way by means of Psychotherapy Process Q Set (PQS) ratings of the transcripts of the sessions.
  •Measures during A phases: Besides the SCID-I (session 1 and 2 of each A phase) and SCID-II (session 3 of each A phase) interviews, the therapist will administer the Depressive Experiences Questionnaire (DEQ).

SECONDARY OUTCOMES:
improvement in relational capacities | 25 weeks
  • Measures that are applied each session (also during A phases): The relational capacities (CDPS-RC) and insight (CDPS-IN) subscales of the Capacity for Dynamic Process Scale (CDPRS) of nine researcher-rated items.
  • Measures that are applied during A phases: The therapist will administer the Clinical Diagnostic Interview (CDI, session 4 and 5 of each A phase),and a broad-spectrum set of self-report outcome measures, including the Symptom Check List (SCL-90-R), the Inventory of Interpersonal Problems - 64 (IIP-64), the SELVES and the Quality of Life Inventory (QOLI).
improvement in insight | 25 weeks
  * Measures that are applied each session (also during A phases): The relational capacities (CDPS-RC) and insight (CDPS-IN) subscales of the Capacity for Dynamic Process Scale (CDPRS) of nine researcher-rated items.
  * Measures that are applied during A phases: The therapist will administer the Clinical Diagnostic Interview (CDI, session 4 and 5 of each A phase),and a broad-spectrum set of self-report outcome measures, including the Symptom Check List (SCL-90-R), the Inventory of Interpersonal Problems - 64 (IIP-64), the SELVES and the Quality of Life Inventory (QOLI).
improvement in quality of life, a broad range of physical and psychological symptoms. | 25 weeks
  Measures that are applied each session (also during A phases): The relational capacities (CDPS-RC) and insight (CDPS-IN) subscales of the Capacity for Dynamic Process Scale (CDPRS) of nine researcher-rated items.
  Measures that are applied during A phases: The therapist will administer the Clinical Diagnostic Interview (CDI, session 4 and 5 of each A phase),and a broad-spectrum set of self-report outcome measures, including the Symptom Check List (SCL-90-R), the Inventory of Interpersonal Problems - 64 (IIP-64), the SELVES and the Quality of Life Inventory (QOLI).

CONTACTS AND LOCATIONS:
Overall Officials: Stijn Vanheule, Prof Phd, Principal Investigator — University Ghent; Gilbert Lemmens, Phd MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University, Ghent, Belgium